CLINICAL TRIAL: NCT01188850
Title: Phase I, Open-label Study to Evaluate the Safety, Tolerability and Immunogenicity of a Fourth Dose of Human Papillomavirus (HPV) DNA Plasmid (VGX-3100) + Electroporation (EP) in Adult Females Previously Immunized With VGX-3100
Brief Title: Fourth Dose of Human Papillomavirus (HPV) DNA Plasmid (VGX-3100) + EP in Adult Females Previously Vaccinated With Three Doses of VGX-3100
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HPV-002
Record Dates: First submitted 2010-08-05; First posted 2010-08-26 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Human Papillomavirus (HPV)
Keywords: CIN 2 or 3; cervical cancer; Human Papillomavirus (HPV)
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — VGX-3100

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 6mg of DNA/dose (Experimental): Subjects who have previously received a 3 dose series of VGX-3100 containing either 0.6, 2 or 6mg DNA/dose will receive a fourth dose of VGX-3100 containing 6mg of DNA/dose administered via IM injection + electroporation at Day 0
  Interventions: Biological: VGX-3100

INTERVENTIONS:
Biological: VGX-3100 — DNA plasmid delivered via IM injection + electroporation using CELLECTRA device

SUMMARY:
DNA vaccines, which are small pieces of DNA also known as plasmids, have several advantages over traditional vaccines such as live attenuated virus and recombinant protein-based vaccines. DNA vaccines appear to be well tolerated in humans. Therefore, the investigators have developed our DNA vaccine, VGX-3100, to include plasmids targeting E6 and E7 proteins of both HPV subtypes 16 and 18. The investigators have chosen to deliver our candidate vaccines via electroporation (EP) using the CELLECTRA constant current device to deliver a small electric charge following intramuscular (IM) injection, since animal studies have shown that this delivery method increases the immune response to our DNA vaccine leading to a decrease in the size of tumors caused by HPV 16 and 18. In study HPV-001, the vaccine was given to subjects with a history of CIN 2 and 3 who had been previously treated by surgery. This study is proposed to vaccinate the same subjects with a fourth dose of the VGX-3100 to determine the safety and immune response.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent in accordance with institutional guidelines;
2. Successful enrollment in and completion of all study procedures and follow-up in study HPV-001.
3. Female 18-46 years of age;
4. Post surgical (including LEEP and conization) or ablative treatment and a diagnosis of CIN 2 or 3, while under physician care as per ASCCP guidelines (Appendix C);
5. Normal ECG and CPK, as judged by Grade 0-1 as per Toxicity Grading Scale for Healthy Adults (Appendix B) done up to 30 days prior to administration of study treatment;
6. Body mass index (BMI) ≤30 kg/m2;
7. Women of child-bearing potential (WOCBP) agree to remain sexually abstinent, use medically effective contraception (oral contraception, barrier methods, spermicide, etc), or have a partner who is sterile (i.e., vasectomy) from enrollment to study discharge;
8. Able and willing to comply with all study procedures.

Exclusion Criteria:

1. Active infection with herpes simplex virus (HSV);
2. Pregnant or breast feeding subjects;
3. Any concurrent condition requiring the continued use of systemic or topical steroids (excluding inhaled and eye drop-containing corticosteroids) or the use of immunosuppressive agents. All other corticosteroids must be discontinued > 4 weeks prior to Day 1 of treatment;
4. Administration of any blood product within 3 months of enrollment;
5. Administration of any vaccine within 6 weeks of enrollment;
6. Patient is currently participating or has participated in a study with an investigational compound or device other than VGX-3100 within 30 days of signing informed consent;
7. Metal implants at the site of injection;
8. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements;
9. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (i.e. infections disease) illness must not be enrolled into this study;
10. Any other conditions judged by the investigator that would limit the evaluation of a subject.

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2010-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10-20 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of a fourth dose of VGX-3100 | through Month 6 (end of study)
  Safety and tolerability of a fourth dose of VGX-3100, administered by IM injection with EP to adult females who have been previously immunized with three doses of VGX-3100

SECONDARY OUTCOMES:
Humoral and cellular immune responses to VGX-3100 | through Month 6 (end of study)
  Humoral and cellular immune responses to VGX-3100 in blood samples obtained from study subjects after a fourth dose of VGX-3100 (6 mg) in adult female subjects who have been previously vaccinated with a three dose series of VGX-3100 containing 0.6, 2 or 6 mg of DNA/dose.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Parker, MD, Principal Investigator — Lyndhurst Gynecologic Associates; John Sunyecz, MD, Principal Investigator — Laurel Highlands, OB/GYN, P.C.; Javier Morales, MD, Principal Investigator — Clinical Research Puerto Rico
Locations (3):
- United States (2):
  - Lyndhurst Gynecologic Associates, Winston-Salem, North Carolina
  - Laurel Highlands, OB/GYN, P.C., Hopwood, Pennsylvania
- Clinical Research Puerto Rico, San Juan, Puerto Rico